CLINICAL TRIAL: NCT06273449
Title: A Smart Digital Workflow Towards High Precision and Through-Put Production for Removable Partial Dentures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Dental Centre, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 385/2023
Record Dates: First submitted 2023-11-07; First posted 2024-02-22 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Partial-edentulism

STUDY DESIGN:
Intervention Model Description: 1. Conventional: The Standard of Care (SOC) workflow, which will act as a baseline compared to the other 2 groups.
  2. Partial digital workflow: Adopts the same teeth profile capture method, where a physical impression of teeth profile is taken from the subject. However, instead of using physical wax pattern on the stone model for design, the stone model is scanned and, on the scan, the design is performed digitally. For fabrication of RPD, instead of using lost wax casting, the digital design is used for additive manufacturing.
  3. SmartRPD digital workflow Adopts a different teeth profile capture method by using the intraoral scanner to digitally scan and save the subject's teeth profile. From the intraoral scan, a digital model of the subject's teeth profile is created but on the digital model instead, the design of RPD is digitally performed. The digital design is used for additive manufacturing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (No Intervention): Conventional:
  The Standard of Care (SOC) workflow, which will act as a baseline compared to the other 2 groups.
  Teeth Profile Capture Method: Physical impression RPD Design Method: Based on stone model, using wax pattern RPD Fabrication Method: Lost wax casting
- Group 2 (Experimental): Partial Digital:
  Similar to the SOC, Group 2 adopts the same teeth profile capture method, where a physical impression of teeth profile is taken from the subject. However, instead of using physical wax pattern on the stone model for design, the stone model is scanned and, on the scan, the design is performed digitally. For fabrication of RPD in Group 2, instead of using lost wax casting as per the SOC, the digital design is used for additive manufacturing.
  Interventions: Device: Group 2 - 3D Printed Removable Partial Denture
- Group 3 (Experimental): SmartRPD Digital:
  Group 3 adopts a different teeth profile capture method by using the intraoral scanner to digitally scan and save the subject's teeth profile. From the intraoral scan, a digital model of the subject's teeth profile is created. Similar to Group 2, but on the digital model instead, the design of RPD is digitally performed. The digital design, as per Group 2, is used for additive manufacturing.
  Interventions: Device: Group 3 - 3D Printed Removable Partial Denture

INTERVENTIONS:
Device: Group 3 - 3D Printed Removable Partial Denture — Teeth Profile Capture Method: Intraoral scan RPD Design Method: Based on intraoral scan, using design software RPD Fabrication Method: Additive manufacturing
  Arms: Group 3
Device: Group 2 - 3D Printed Removable Partial Denture — Teeth Profile Capture Method: Physical impression RPD Design Method: Based on stone model, using design software RPD Fabrication Method: Additive manufacturing
  Arms: Group 2

SUMMARY:
Tooth loss is a major chronic problem in dentistry and edentulous elderly endures poorer quality of life worldwide. Removable partial dentures (RPDs) are the most widely accepted and cost-effective treatment for patients to restore oral functions. RPDs contain three components including the metal framework, denture base and acrylic teeth. Conventionally, RPD fabrication involves tedious clinical and dental laboratory procedures and is time consuming, labour-intensive, and often imprecise, therefore incapable of meeting the growing demands of RPD by an ageing population. The challenges to achieve a high quality and high-throughput RPD service lie in three aspects: 1) accuracy in capturing oral profile; 2) immediate oral information analysis and device design, and 3) automation in production.

DETAILED DESCRIPTION:
Tooth loss is a major chronic problem in dentistry and edentulous elderly endures poorer quality of life worldwide. Removable partial dentures (RPDs) are the most widely accepted and cost-effective treatment for patients to restore oral functions. RPDs contain three components including the metal framework, denture base and acrylic teeth. Conventionally, RPD fabrication involves tedious clinical and dental laboratory procedures and is time consuming, labour-intensive, and often imprecise, therefore incapable of meeting the growing demands of RPD by an ageing population. The challenges to achieve a high quality and high-throughput RPD service lie in three aspects: 1) accuracy in capturing oral profile; 2) immediate oral information analysis and device design, and 3) automation in production.

Towards this goal, we have developed an intelligent RPD design software prototype, SmartRPD, to generate RPD metal framework design using digital scans from patients. SmartRPD processes patient-specific scanned geometry instantly, provide diagnosis analysis and generate the first draft of metal framework design automatically, powered by a teeth geometry segmentation system, knowledge-based design algorithm and 3D geometry engines. Dentists make the final clinical changes and confirmation before sending the 3D digital files for 3D printing. Thereafter, an altered digital scan technique is used to register a precise digital scan of soft tissues under functioning, using the metal framework as a loading impression tray and digitally align to the initial oral scan. This resulted modified master scan file leads to a more accurate setting for the denture base in the subsequent procedures.

ELIGIBILITY:
Inclusion Criteria:

* above the age of 21 years' old
* medically fit
* with prior denture experience
* either maxillary or mandible partial dentate
* partial edentulism with stable occlusion

Exclusion Criteria:

* History of maladaptation to denture use
* With maxillofacial or mandible bone defect(s)
* Known allergic reaction to cobalt chromium metal

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Precision in Fabricated Metal Frameworks Across Three Workflows | Assessed at the end of the study period, up to 14 months
  The precision of fabricated RPD metal frameworks will be assessed by measuring the gaps between occlusal rests and corresponding rest seats of abutment teeth during the clinical try-in stage. Clinical parameters including support, retention, and stability will be evaluated by calibrated clinical evaluators to compare framework quality among three patient groups.
  Measurement: Gap measurements between occlusal rest and corresponding rest seat
Comparison of Patient Satisfaction with RPD Prostheses Fabricated Using Three Workflows | From date of randomization during first visit till 3rd follow up visit, assessed up to 14 months
  Patient satisfaction with final RPD prostheses will be compared among three workflows. Assessment of patient satisfaction with various oral functions will be conducted using validated denture and oral health impact (OHIP) questionnaires.
  Measurement: Patient-reported satisfaction scores on denture and oral health impact questionnaires.
Comparison of Fabrication Cost and Time Across Three Workflows | Assessed at the end of the study period, up to 14 months
  he study aims to compare fabrication cost and time spent on three workflows. Direct and indirect costs, clinical chair time, and laboratory work time will be measured based on an operational model in a dental clinic. Additionally, exploratory analysis will be conducted to assess changes in quality-adjusted life years attributable to different dental workflows.
  Measurement: Direct and indirect costs, clinical chair time, laboratory work time, and potential changes in quality-adjusted life years.

CONTACTS AND LOCATIONS:
Locations (1):
- National Dental Centre Singapore, Singapore, Singapore